CLINICAL TRIAL: NCT01780220
Title: Safety and Efficacy of Radiotherapy Combined With a 6-month LH-RH Agonist and Abiraterone Hormone Therapy Treatment in Biochemically-relapsing Prostate Cancer Following Surgery
Brief Title: Radiotherapy Plus Hormone Therapy in Biochemically-relapsing Prostate Cancer Patients Following Surgery
Acronym: CARLHA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEP12-UC-0101/1104; 2011-004831-30 (EudraCT Number)
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Biochemically-relapsing Prostate Adenocarcinoma Following Radical Prostatectomy
Keywords: abiraterone; biochemically-relapsing; prostate adenocarcinoma
MeSH Terms: interventions — abiraterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- abiraterone (Experimental): Abiraterone acetate (three dose levels in phase I) + prednisone (10mg/day)+LHRH + Radiotherapy
  Interventions: Drug: Abiraterone

INTERVENTIONS:
Drug: Abiraterone — Abiraterone acetate 1000mg/day + prednisone alone for one month before initiating the sequence of radiotherapy

SUMMARY:
As there is no prospective data on the combination of abiraterone and salvage radiotherapy, the aim of this study is to further evaluate the safety profile of abiraterone acetate plus prednisone in patients with prostate cancer who are biochemically relapsing after surgery and undergo salvage radiotherapy with 6-months LH-RH agonist.

The investigators hypothesize that the toxicity profile of both treatments should not potentiate each other. This study will also provide preliminary data on the efficacy of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed prostate adenocarcinoma
2. The patients should have undergone only surgery for localized prostate adenocarcinoma: pT2, pT3 or pT4 with bladder neck involvement
3. pN0: negative lymphadenectomy at the time of prostatectomy
4. At inclusion the patients should have no clinical signs of progressive disease and should be M0 (bone and pelvic scans).
5. ≥ 18 years of age with life expectancy ≥ 10 years
6. Performance Status (ECOG) ≤ 1
7. PSA ≤ 0.1 ng/ml after prostatectomy (dosage performed within 2 months after surgery)
8. PSA ≥ 0.2 ng/ml et ≤ 2 ng/ml at the time of inclusion
9. Elevation of PSA over three consecutive assays performed in the same laboratory, with a minimal interval of two months between assays, (PSA nadir level followed by two other progressive assays)
10. At least 6 months between surgery and biochemical relapse
11. Serum potassium ≥ 3.5 mmol/L in the 72 hours before first dose of abiraterone acetate
12. Serum creatinine < 1.5 x ULN or a calculated creatinine clearance ≥ 60 mL/min
13. Liver function:

    Serum bilirubin < 1.5 x ULN (except for patients with documented Gilbert's disease) AST and ALT < 2.5 x ULN
14. Patients must be affiliated to a Social Security System.
15. Patient information and written informed consent form signed for both principal and additional research
16. Patients must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

1. pN1: histologically-proven lymph node involvement at initial lymphadenectomy
2. Histology other than adenocarcinoma
3. Previous hormone therapy including prior therapy with ketoconazole or other CYP17 inhibitor(s) for prostate cancer.
4. Patients being treated within the last 14 days prior to inclusion with drugs recognized as being strong inhibitors or inducers of the isoenzyme CYP3A4 (Clarithromycin, Ketoconazole, Itraconazole, Voriconazole, Ritanovir, see appendix 11) or requiring those treatments during the study
5. Active or symptomatic viral hepatitis or chronic liver disease
6. Surgical or chemical castration
7. History of cancer, with the exception of basal cell carcinoma or any other cancer treated in the 5 years before inclusion and in complete remission.
8. Previous pelvic radiotherapy
9. Uncontrolled hypertension (defined as systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive therapy (see appendix 10 for mandatory BP measurement guidelines)
10. Severe and moderate hepatic impairment (Child-Pugh class B and C)
11. Patients with severe and/or uncontrolled medical disease which could compromise participation in the study, such as, but not limited to:

    Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, or New York Heart Association (NYHA) Class III or IV heart disease or cardiac ejection fraction measurement of < 50 % at baseline
12. Known hypersensitivity to any of the study drugs or excipients.
13. Galactosemia, Glucose-galactose malabsorption or lactase deficiency
14. Patients with any psychological, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
15. Individual deprived of liberty or placed under the authority of a tutor.
16. Patients already included in another therapeutic trial with an experimental drug or having been given an experimental drug within a period of 30 days.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
to determine the maximum tolerated dose and the phase II recommended dose of abiraterone acetate treatment plus prednisone and LH-RH agonist combined with prostate radiotherapy | within 11 weeks after Radiotherapy initiation

SECONDARY OUTCOMES:
To evaluate the 3-year biochemical relapse-free survival | 3 years

OTHER OUTCOMES:
overall safety profile | 3 years

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Institut de Cancérologie de l'ouest/René Gauducheau, Saint-Herblain